CLINICAL TRIAL: NCT04989764
Title: COMPARATIVE EFFECTS OF PERIOPERATIVE AND ADJUVANT CHEMOTHERAPY ON OUTCOMES OF OPERABLE GASTRIC CANCER: EXPERIENCE FROM A CANCER CARE CENTER
Status: Completed | Type: Observational
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: EX-05-03-20-40
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer, Outcomes, Pakistan, Adjuvant Chemotherapy, Perioperative Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- perioperative chemotherapy vs. adjuvant therapy in gastric ca patients
- perioperative chemotherapy group vs. adjuvant chemotherapy group

SUMMARY:
* Patients with gastric adenocarcinoma
* Comparison: perioperative chemotherapy vs. adjuvant therapy.
* Sample size differences between the two groups.
* Kaplan meier survival analysis, overall survival and disease free survival

ELIGIBILITY:
Inclusion Criteria:

* We included histologically proven gastric adenocarcinoma patient with operable disease and the patients who completed their prescribed perioperative or adjuvant chemotherapy cycles

Exclusion Criteria:

* Patients were excluded if they had Tis or T1, N0 disease, inoperable disease, metastatic. In addition, all those who did not undergo adequate lymphadenectomy (< D2) or had R1 margins following surgery were excluded

Age Groups: Child, Adult, Older Adult
Study Population: cancer patients who had histologically proven gastric adenocarcinoma diagnosed at Shaukat Khanum Memorial Cancer Hospital and Research Centre (SKMCH & RC), between January 2015 and December 2019
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
The overall survival | from January 2015 till December 2019
  The overall survival (OS) was defined as the length of the time from date of diagnosis till last follow-up or death
The disease-free survival | from January 2015 till December 2019
  The disease free survival (DFS) as the length of the time from date of last treatment which is either perioperative or adjuvant chemotherapy to tumor relapse or death.

IPD SHARING:
Plan to Share IPD: Undecided